CLINICAL TRIAL: NCT00638365
Title: A Phase I/II Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose Escalation Study of KB001 in Cystic Fibrosis Patients Infected With Pseudomonas Aeruginosa
Brief Title: Dose Escalation Study of KB001 in Cystic Fibrosis Patients Infected With Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB001-03
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2011-08-08 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, Pseudomonas aeruginosa, Pulmonary CF
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): KB001, a monoclonal antibody
  Interventions: Biological: KB001
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: KB001 — Single-dose, 3mg/kg or 10mg/kg dose administered intravenously
  Other Names: KB001-recombinant human anti-Pa PcrV Fab antibody
  Arms: 1
Other: Placebo — Placebo single-dose administered intravenously
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a single dose of KB001 in Cystic Fibrosis patients infected with Pseudomonas aeruginosa (Pa)

DETAILED DESCRIPTION:
CF patients often have lung infections. Pseudomonas aeruginosa (Pa) is the most significant bacteria in CF, with up to 80% of CF patients eventually becoming infected. These patients are often treated with antibiotics with variable results. This study will examine the impact of a single-dose of an investigational drug, KB001, on Pa bacteria in the CF lung.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Confirmed diagnosis of CF based on the following criteria:

Positive sweat chloride greater than 60mEq/liter, and/or a genotype with 2 identifiable mutations consistent with CF, and one or more clinical features consistent with the CF phenotype

* Age >/= 18 years of age with the potential for age 12 >/=
* Screening Pa sputum culture
* FEV1% predicted >/= 40 (based on Wang's equations for Males aged 12-17 and females 12-15 years, and Hankinson's equations for all other patients)

Exclusion Criteria:

* Evidence of an acute respiratory infection or pulmonary exacerbation within 4 weeks prior to day 0
* Use of systemic corticosteroids or antibiotics within 4 weeks prior to day 0, or cyclic inhaled antibiotics within 14 days prior to day 0.
* History of positive B. cepacia complex, organ transplantation, hepatic disease or venal dysfunction
* Current cigarette smoker, history of drug addiction or alcohol abuse
* Use of investigational medication or participation in an investigational study within 4 weeks prior to day 0
* Women who are pregnant or breastfeeding and patients and/or partner unwilling to use an effective form of barrier contraception throughout the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Milla, MD, Principal Investigator — Stanford University; Nestor A. Molfino, MD, MSc, Study Director — Humanigen, Inc.
Locations (11):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Lucille Packard Children's Hospital at Stanford, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Milla CE, Chmiel JF, Accurso FJ, VanDevanter DR, Konstan MW, Yarranton G, Geller DE; KB001 Study Group. Anti-PcrV antibody in cystic fibrosis: a novel approach targeting Pseudomonas aeruginosa airway infection. Pediatr Pulmonol. 2014 Jul;49(7):650-8. doi: 10.1002/ppul.22890. Epub 2013 Sep 9. PMID 24019259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, randomized, double-blind, placebo-controlled safety and PK study.
Pre-assignment Details: Two cohorts of subjects were randomized 2:1 and received a single intravenous (IV) infusion of KB001 or Placebo. Cohort 1 received KB001 at 3 mg/kg. Cohort 2 was enrolled at 10 mg/kg. The Placebo groups were combined for analysis.
Period: Overall Study
Arm/Group | Placebo | KB001, 3 mg/kg | KB001, 10 mg/kg
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | KB001, 3 mg/kg | KB001, 10 mg/kg | Total
Number analyzed (Participants) | 9 | 10 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 0 | 2
  Between 18 and 65 years | 9 | 8 | 8 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 2 | 9
  Male | 7 | 5 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of a Single-dose of KB001.
Description: Safety assessments were conducted after completion of day 28. AEs were followed through completion of day 56.
Time Frame: Day 28
Population: Safety population: all subjects randomized and receiving any study medication.
Measure: Number; unit: Number of participants experiencing AEs
Arm/Group | Placebo | KB001, 3 mg/kg | KB001, 10 mg/kg
Number analyzed (Participants) | 9 | 10 | 8
Number of participants experiencing AEs | 7 | 10 | 8

ADVERSE EVENTS:
Time Frame: 56 Days
Arm/Group | Placebo | KB001, 3 mg/kg | KB001, 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 7/9 | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | KB001, 3 mg/kg (N=10) | KB001, 10 mg/kg (N=8)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | KB001, 3 mg/kg (N=10) | KB001, 10 mg/kg (N=8)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Stomach pain
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Exacerbation of asthma
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Breath Sounds Abnormal (Investigations) | 2 (2) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Angular stromatitis
Chest Discomfort (General disorders) | 0 (0) | 2 (2) | 2 (2) — Chest soreness
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Crepitations (General disorders) | 0 (0) | 0 (0) | 1 (2)
Cystic Fibrosis Lung (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) — Cystic Fibrosis pumonary exacerbation
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Hoarse voice
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) — Shortness of breath
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Forced Expiratory Volume Decreased (Investigations) | 0 (0) | 4 (6) | 0 (0)
Haemoptysis (hemoptysis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4) — Intermittent headache
Heart Rate Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Infusion Related Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) — Adverse infusion reaction
Infusion Site Discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Rash (General disorders) | 1 (1) | 0 (0) | 1 (1) — Faint scattered erythematous macules at prior infusion site
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) — Increased nasal congestion
Nausea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — Nausea
Oral Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pancreatitis, mild
Pharyngolaryingeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Sore throat
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Mouth pain from wisdom tooth extraction
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) — Increased sputum production
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Feet itching
Pyrexia (fever) (General disorders) | 1 (1) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Chest congestion
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Runny nose
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Sinus Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — Sinus infection
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Itchy throat
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — Patient hears ear clicking
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Urticaria right anterior abdomen
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has right of first publication of trial results, which will be a joint, multi-center publication of the study results from all appropriate sites contributing data, analysis and comments.